CLINICAL TRIAL: NCT05117996
Title: Simplified Bowel Preparation Versus Standard Bowel Preparation Before Capsule Endoscopy in Patients With Crohn's Disease: a Prospective Randomized Controlled Multicenter Study
Brief Title: Simplified Bowel Preparation Versus Standard Bowel Preparation Before Capsule Endoscopy in Patients With Crohn's Disease
Acronym: CROHN-PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC21_0123
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard small bowel preparation (Active Comparator): 2 L of polyethylene glycol and free residue diet the day before the capsule endoscopy. 2 mL of Babyspasmyl after ingestion of capsule
  Interventions: Other: capsule endoscopy; Other: standard small bowel preparation
- Simplified small bowel preparation (Experimental): Liquid diet the evening before and water on the morning of the capsule endoscopy. 2 mL of Babyspasmyl after ingestion of capsule
  Interventions: Other: capsule endoscopy; Other: Simplified small bowel preparation

INTERVENTIONS:
Other: capsule endoscopy — capsule endoscopy
Other: standard small bowel preparation — 2 L of polyethylene glycol and free residue diet the day before the capsule endoscopy. 2 mL of Babyspasmyl after ingestion of capsule
  Arms: Standard small bowel preparation
Other: Simplified small bowel preparation — Liquid diet the evening before and water on the morning of the capsule endoscopy. 2 mL of Babyspasmyl after ingestion of capsule
  Arms: Simplified small bowel preparation

SUMMARY:
The European guidelines currently recommend to use 2 L of polyethylene glycol and free residue diet before any capsule endoscopy. However, up to now, no studies have been conducted to specifically evaluate bowel preparation modalities before small bowel capsule endoscopy in patients with Crohn's disease.

In patients with Crohn's disease and small bowel ulcers, polyethylene glycol may remove some fibrin from these ulcers and alter bowel preparation. Moreover, it is important to select the most acceptable bowel preparation because patients with Crohn's disease will have to repeat capsule endoscopy several times after initiating treatment, for monitoring under treatment, or for detection of post-operative recurrence.

In a preliminary retrospective study, it has been suggested that a simplified bowel preparation with liquid diet the evening before and water on the morning of the capsule endoscopy induced a better bowel preparation than the standard method with polyethylene glycol.

Thus, the aim of the study is to demonstrate the superiority of this simplified bowel preparation compared to the standard preparation modality in terms of quality of bowel preparation, patient's acceptability and diagnostic yield.

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory bowel disease characterized by the presence of ulcers that can affect the entire digestive tract, from the mouth to the anus. The existence of small bowel lesions is pejorative and associated with poorer outcomes and a higher risk of intestinal resection.

Small bowel capsule endoscopy allows the visualization of the entire small bowel in a non-invasive and outpatient setting, without any anesthesia. It is the exam with the best diagnostic yield for the detection of small bowel ulcers in patients with Crohn's disease. Moreover, it allows the monitoring of patients after initiating treatment to assess mucosal healing and the detection of post-operative recurrence.

As for any endoscopic examinations, its acceptability depends on bowel preparation modalities. The European Society of Gastrointestinal Endoscopy (ESGE) currently recommends to use 2 L of polyethylene glycol and free residue diet before any capsule endoscopy. However, patients with Crohn's disease were a minority (< 1.5 %) in the studies on which these guidelines are based on.

Yet, in patients with small bowel Crohn's disease, polyethylene glycol may remove some fibrin from the ulcers and hence, alter bowel preparation. Moreover, it is important to select the most acceptable bowel preparation because patients with Crohn's disease will have to repeat capsule endoscopy several times after initiating treatment, for monitoring under treatment, or for detection of post-operative recurrence.

A preliminary retrospective study suggested that a simplified bowel preparation with liquid diet the evening before and water on the morning of the capsule endoscopy induced a better bowel preparation than the standard method with polyethylene glycol.

Thus, the aim of CROHN-PREP study is to demonstrate the superiority of this simplified bowel preparation compared to the standard preparation modality in terms of quality of bowel preparation, patient's acceptability and diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged over 18 years old
* With an established diagnosis of Crohn's disease, whether active or quiescent
* With an indication of a small bowel capsule endoscopy
* Without any small bowel stricture (patency capsule procedure on the 7 days before the capsule endoscopy)
* Registered with a social security scheme
* Having provided their oral consent for the study after appropriate information

Exclusion Criteria:

* - Patients aged below 18 years old
* Diagnosis of ulcerative colitis or IBD unclassified
* Presence of an ileostomy
* Presence of a small bowel syndrome
* Symptoms suggestive of a small bowel stricture
* Retention of the patency capsule on an abdominal X-ray performed 48 hours after the ingestion
* Abdominal pain after the ingestion of the patency capsule
* Planned abdominal surgery in the next month
* Known intestinal fistula
* Swallowing disorders
* Established diagnosis of delayed gastric emptying or suggestive symptoms
* Intake of non-steroidal anti-inflammatory drugs (NSAIDs) in the month prior to the capsule endoscopy
* Intake of oral iron supplementation in the week prior to the capsule endoscopy
* Intake of oral 5-ASA granules in the week prior to the capsule endoscopy
* Ongoing pregnancy
* Presence of a pace-maker or implantable defibrillator
* Known allergy to polyethylene glycol or to lactose
* Vulnerable people i.e. adults under a legal protection regime (guardianship, trusteeship, judicial safeguard)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
KODA score (entire small bowel) | through the reading of the capsule endoscopy, an average of 6 months
  Small bowel preparation quality (entire small bowel)

SECONDARY OUTCOMES:
KODA score for each small bowel segment | through the reading of the capsule endoscopy, an average of 6 months
  Small bowel preparation quality (by segment : upper/middle/lower third)
Qualitative assessment by the reader | through the reading of the capsule endoscopy, an average of 6 months
  Proportion of images in which preparation is considered as "good", "moderate" or "low" by the reader (by segment)
Quantitative assessment of acceptability of preparation | Immediately before the capsule endoscopy
  Patient's acceptability of the bowel preparation on a visual analog scale between 0 (nil) to 10 (excellent)
Quantitative assessment on a visual analog scale between 0 (nil) to 10 (excellent) | Immediately before the capsule endoscopy
  Patient's acceptability of the examination on a visual analog scale between 0 (nil) to 10 (excellent)
Lewis score | through the reading of the capsule endoscopy, an average of 6 months
  Diagnostic yield evaluation
complete examinations | through the reading of the capsule endoscopy, an average of 6 months
  Percentage of complete examinations defined by the visualization of the first duodenal image and the first caecal image
Small bowel transit time | through the reading of the capsule endoscopy, an average of 6 months
  Recording time between the visualization of the first duodenal image and the first caecal image, if visualized

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Angers University Hospital, Angers
  - Vendée departmental hospital, La Roche-sur-Yon
  - Clinique Jules Verne, Nantes
  - Hopital privé Confluent, Nantes
  - Nantes University Hospital, Nantes
  - Rennes University hospital, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rouveyre R, Coudol S, Collins M, de Maissin A, Flamant M, Trang C, Freyssinet M, Bouguen G, Dib N, Bourreille A, Le Berre C. Clinical Trial: Simplified Bowel Preparation for Small Bowel Capsule Endoscopy in Crohn's Disease. Aliment Pharmacol Ther. 2026 Jan;63(1):57-69. doi: 10.1111/apt.70417. Epub 2025 Oct 20. PMID 41116605